CLINICAL TRIAL: NCT05355246
Title: Effects of Assisted Sit-up Exercise Versus Swiss Ball Pikes on Pain and Disability in Patients With Postpartum Low Back Pain.
Brief Title: Effects of Assisted Sit-up Exercise vs Swiss Ball Pikes on Postpartum Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0503 Romaisa
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Postpartum Disorder; Lumbar Pain Syndrome; Activation, Patient
MeSH Terms: conditions — Puerperal Disorders; Somatoform Disorders; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- assisted sit-up exercises Group (Experimental): Group A patients will be instructed to perform assisted sit-up exercises by lying on their back and lifting their torso. They will use their body weight to strengthen and tone the core stabilizing abdominal muscles. This exercise will perform a minimum of five and a maximum of 10 repetitions, two times a day and two days a week.
  Interventions: Other: assisted sit-up exercises
- swiss ball pikes exercises Group (Active Comparator): Group B patients will be instructed to perform swiss ball pikes by getting into the pushup position, the rest of the tops of their feet on a swiss ball. Each patient should keep her legs as straight as possible, bend their hips and try to pull their feet towards their chest so that the ball rolls forward. Hold at the top for three to four seconds, then slowly roll back to the starting position. This exercise will perform a minimum of one or two and a maximum of 10 repetitions, two times a day and two days a week. Both exercises will be performed for 12 weeks in both groups.
  Interventions: Other: swiss ball pikes exercises

INTERVENTIONS:
Other: assisted sit-up exercises — Group A patients will be instructed to perform assisted sit-up exercises by lying on their back and lifting their torso. They will use their body weight to strengthen and tone the core stabilizing abdominal muscles. This exercise will perform a minimum of five and maximum of 10 repetitions, two times a day and two days a week. Isometrics, back stretching, and strengthening exercises will be given as a common intervention for both groups before starting treatment session.
  Arms: assisted sit-up exercises Group
Other: swiss ball pikes exercises — Group B patients will be instructed to perform swiss ball pikes by getting into the pushup position, the rest of the tops of their feet on a swiss ball. Each patient should keep her legs as straight as possible, bend her hips and try to pull her feet towards their chest so that the ball rolls forward. Hold at the top for three to four seconds, then slowly roll back to the starting position. This exercise will perform a minimum of one or two and a maximum of 10 repetitions, two times a day and two days a week. Both exercises will be performed for 12 weeks in both groups. Isometrics, back stretching, and strengthening exercises will be given as a common intervention for both groups before starting the treatment session.
  Arms: swiss ball pikes exercises Group

SUMMARY:
The aim of this study is to evaluate and compare the effectiveness of assisted sit-up exercise and swiss ball pikes on the treatment of pain and disability of postpartum low back pain. The current study will compare the use of assisted sit-up exercise and swiss ball pikes. The current study is novel in a way that there is limited literature about treating postpartum low back pain with physical strengthening exercises. These two methods will be employed to see if they improve ranges along with accompanying pain and disability.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial. Subjects with postpartum low back pain meeting the predetermined inclusion and exclusion criteria will divide into two groups. Pre-assessment will be done using the Numeric Pain Rating Scale & Roland-Morris Questionnaire as subjective measurements. Subjects in one group will be treated with assisted sit-up exercise and the other will be treated with swiss ball pikes. Each subject will receive a total of 12 treatment sessions, with 2 treatment sessions per week. Post-treatment reading for numeric pain rating scale and Roland-Morris questionnaire will be recorded after the end of the 4th, 8th, and 12th treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 40 years.
* Back pain without leg pain for at least three months postpartum period.
* Pain intensity of numeric pain rating scale ranges between 6 to 10.
* Intensity of pain limited daily work activities.

Exclusion Criteria:

* Any kind of infection, malignancy, inflammation, and structural deformity present in the lumbar and pelvic region.
* Neurologic signs
* Trauma history of the lumbar and pelvic region
* Any lumber or abdominal surgery
* Pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | up to 6 weeks
  An outcome measure that is a segmented numeric version of visual analogue scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of patient's pain. The common format is horizontal bar or line and NPRS is anchored by terms describing pain and severity extremes.
Ronald Morris Disability (RMD) questionnaire | up to 6 weeks
  a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. This questionnaire has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ha VVA, Zhao Y, Pham MN, Binns CW, Nguyen CL, Nguyen PTH, Chu TK, Lee AH. Physical Activity During Pregnancy and Postpartum Low Back Pain: A Prospective Cohort Study in Vietnam. Asia Pac J Public Health. 2019 Nov;31(8):701-709. doi: 10.1177/1010539519890148. PMID 31852228
- [Background] Li YP, Cui X, Liu SC, Zhang SH, Zhao YH. Neuromuscular electrical stimulation for treating postpartum low back pain. Medicine (Baltimore). 2018 Jul;97(28):e11426. doi: 10.1097/MD.0000000000011426. PMID 29995793
- [Background] Tavares P, Barrett J, Hogg-Johnson S, Ho S, Corso M, Batley S, Wishloff K, Weis CA. Prevalence of Low Back Pain, Pelvic Girdle Pain, and Combination Pain in a Postpartum Ontario Population. J Obstet Gynaecol Can. 2020 Apr;42(4):473-480. doi: 10.1016/j.jogc.2019.08.030. Epub 2019 Dec 18. PMID 31864910
- [Background] Ehsani F, Sahebi N, Shanbehzadeh S, Arab AM, ShahAli S. Stabilization exercise affects function of transverse abdominis and pelvic floor muscles in women with postpartum lumbo-pelvic pain: a double-blinded randomized clinical trial study. Int Urogynecol J. 2020 Jan;31(1):197-204. doi: 10.1007/s00192-019-03877-1. Epub 2019 Apr 23. PMID 31016337
- [Background] Hu X, Ma M, Zhao X, Sun W, Liu Y, Zheng Z, Xu L. Effects of exercise therapy for pregnancy-related low back pain and pelvic pain: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Jan;99(3):e17318. doi: 10.1097/MD.0000000000017318. PMID 32011431
- [Background] Rathore Vs. effect of swiss ball training on breath holding capacity of male physical education students.
- [Background] Bae CR, Jin Y, Yoon BC, Kim NH, Park KW, Lee SH. Effects of assisted sit-up exercise compared to core stabilization exercise on patients with non-specific low back pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018;31(5):871-880. doi: 10.3233/BMR-170997. PMID 29889057
- [Background] Escamilla RF, Lewis C, Bell D, Bramblet G, Daffron J, Lambert S, Pecson A, Imamura R, Paulos L, Andrews JR. Core muscle activation during Swiss ball and traditional abdominal exercises. J Orthop Sports Phys Ther. 2010 May;40(5):265-76. doi: 10.2519/jospt.2010.3073. PMID 20436242
- [Background] Cheng HY, Carol S, Wu B, Cheng YF. Effect of acupressure on postpartum low back pain, salivary cortisol, physical limitations, and depression: a randomized controlled pilot study. J Tradit Chin Med. 2020 Feb;40(1):128-136. PMID 32227774